CLINICAL TRIAL: NCT04705779
Title: The HARMONY Study: A Culturally-relevant, Randomized-controlled, Stress Management Intervention to Reduce Cardiometabolic Risk in African American Women
Brief Title: The HARMONY Study: A Intervention to Reduce Cardiometabolic Risk in African American Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 20-2193; 1R01MD015388-01A1 (NIH)
Record Dates: First submitted 2021-01-08; First posted 2021-01-12 (Actual); Results first posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-03

CONDITIONS: Heart Diseases; Stroke; Pre-diabetes; Hypertension; Obesity; Overweight; Stress
Keywords: HARMONY
MeSH Terms: conditions — Heart Diseases; Stroke; Glucose Intolerance; Hypertension; Obesity; Overweight | interventions — Harmony Hard; Nutritional Status

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HARMONY (Experimental): Following screening, participation includes 8 regular sessions occurring over 4 months followed by 6 monthly booster sessions. Overall, study participation will last approximately 14 months.
  Interventions: Behavioral: HARMONY
- Nutrition and Exercise Education Workgroup (NEEW) (Active Comparator): Following screening, participation includes 8 regular sessions occurring over 4 months followed by 6 monthly booster sessions. Overall, study participation will last approximately 14 months.
  Interventions: Behavioral: Nutrition and Exercise Education (NEEW)

INTERVENTIONS:
Behavioral: HARMONY — The HARMONY intervention will be delivered over 8 every-other-week sessions and 6 monthly booster sessions. Each session will have three components; an exercise sampler, cool down and tailored education on cardiometabolic prevention and risk reductions.
  Arms: HARMONY
Behavioral: Nutrition and Exercise Education (NEEW) — The Nutrition and Exercise Workgroup (NEEW) group will be delivered over 8 every-other-week sessions and 6 monthly booster sessions. Each session will have three components; an exercise sampler, cool down and tailored education on cardiometabolic prevention and risk reductions.
  Arms: Nutrition and Exercise Education Workgroup (NEEW)

SUMMARY:
This study will test whether a culturally-tailored nutrition and exercise intervention designed for African-American women will lead to sustained improvements in exercise and healthy eating through improvements in self-management mediators: mindfulness, stress management, positive reappraisal, self-regulation, and self-efficacy.

DETAILED DESCRIPTION:
Among all groups of women in the US, African American women (AAW) have the highest rates of death and disability from chronic cardiometabolic (CM) illnesses. Furthermore, AAW have inadequate engagement in exercise and are least successful at achieving and sustaining CM risk-reduction goals compared to all men and women of other racial/ethnic groups, despite participating in comprehensive lifestyle interventions. These alarming disparities are due in part to disproportionately high rates of psychological stress. A shortcoming of interventions with AAW is an inadequate focus on stress exposure, including gender and racialized stress, stress physiology, and stress-related barriers to healthy eating and exercise to reduce CM risk. In response, the HARMONY study is a randomized controlled trial to test a culturally-tailored nutrition and exercise intervention to manage stress, designed to help AAW build on their strengths to promote self-management and to reduce stress-related CM risk. Certain information about the interventions is not disclosed to protect the scientific integrity of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported African American or Black woman
* BMI= 25-39 kg/m^2 (confirmed at baseline assessment)
* At least one cardiometabolic risk factor:
* < 150 minutes of self-reported moderate to vigorous exercise
* History of gestational diabetes
* Parent or sibling with prediabetes or diabetes
* Personal or family history of hypertension (=130/80)
* Prediabetes or impaired glucose metabolism (HgbA1c 5.7-6.5)
* Personal or family history of abnormal cholesterol levels
* At least 18 years of age
* Able to read/speak English
* Willing to attend scheduled classes, complete internet surveys and biomarker assessments
* Able/willing to engage in moderate to vigorous exercise
* Ambulatory
* Superwoman Schema Questionnaire score indicating at least moderate endorsement of one or more subscales (strength: 7; motional suppression: 7; resistance of vulnerability: 8; motivation to succeed: 7; or helping others: 10) or a total score of 20 or greater
* A Perceived Stress Scale-14 score of >5 or self-report at least "some" general stress.

Exclusion Criteria:

* Pregnant/anticipated pregnancy
* Substance use, mental health or medical condition that will prevent the ability to participate in the intervention
* Use of weight loss medication
* Current or recent (<6 months prior to enrollment) engagement in another weight loss or meditation program
* Impaired cognition (inability to follow and respond appropriately during screening).
* Diabetes diagnosis
* Has a confirmed BMI lower than 25 or higher than 39
* Does not have access to a smartphone or computer with internet access
* Lives in the same household as someone who is currently in the study or was previously in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2025-02-07 (Actual); Study Completion 2025-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Giscombe, PhD, RN, PMHNP-BC, FAAN, Principal Investigator — The University of North Carolina at Chapel Hill, School of Nursing
Locations (1):
- The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared up to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Time Frame: The data will become available per NIH policy, which is no later than the acceptance for publication of the main findings from the dataset.
Access Criteria: All researchers who desire to access the individual participant data must enter into a data-sharing agreement.

REFERENCES:
- [Derived] Woods-Giscombe CL, Gaylord S, Bradford A, Vines S, Eason K, Smith R, Addo-Mensah D, Lackey C, Dsouza V, Sheffield-Abdullah K, Day T, Green-Scott K, Chilcoat A, Peace-Coard A, Chalmers L, Evenson KR, Samuel-Hodge C, Lewis TT, Crandell J, Corbie G, Faurot K. Protocol of the HARMONY study: A culturally relevant, randomized-controlled, stress management intervention to reduce cardiometabolic risk in African American women. Contemp Clin Trials. 2024 Nov;146:107604. doi: 10.1016/j.cct.2024.107604. Epub 2024 Jun 10. PMID 38866096

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 175 participants who signed informed consent, 173 started the study and received an intervention.
Period: Overall Study
Arm/Group | HARMONY | Nutrition and Exercise Education Workgroup (NEEW)
Started | 87 | 86
Completed | 49 | 43
Not Completed | 38 | 43

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HARMONY | Nutrition and Exercise Education Workgroup (NEEW) | Total
Number analyzed (Participants) | 87 | 86 | 173
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.8 (15.2) | 48.6 (14.6) | 49.2 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 86 | 173
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black and Non-Hispanic | 72 | 71 | 143
  Black and Hispanic | 5 | 2 | 7
  African and Non-Hispanic | 2 | 4 | 6
  Black and West Indian or Caribbean, and Non-Hispanic | 4 | 4 | 8
  Black and African, and Non-Hispanic | 3 | 0 | 3
  Black and West Indian or Caribbean and Native American, and Non-Hispanic | 0 | 1 | 1
  Black and Native American ,Black and West Indian or Caribbean, and Non-Hispanic | 1 | 3 | 4
  Black, Native American, and Creole, and Non-Hispanic | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 87 | 86 | 173

OUTCOME MEASURES:

1. Primary Outcome: Change in Amount of Moderate to Vigorous Physical Activity
Description: The participant's moderate to vigorous physical activity will be measured by triaxial accelerometry. Participants are instructed to wear the accelerometer for seven full days; the average number of minutes of MVPA per 24-hour period is computed. Results will be reported in minutes per day.
Time Frame: Baseline, 48 weeks after first group session
Population: Participants who wore the accelerometer for at least 8 hours at each timepoint.
Measure: Mean (Standard Deviation); unit: minutes/day
Arm/Group | HARMONY | Nutrition and Exercise Education Workgroup (NEEW)
Number analyzed (Participants) | 41 | 33
minutes/day | -5.89 (63.56) | -11.24 (58.40)

2. Primary Outcome: Change in the Dietary Risk Assessment Score
Description: The participant's dietary intake will be assessed using the dietary risk assessment, which includes 54 items. The dietary risk assessment measures the healthiness of a participant's eating habits. Score ranges from 0 to 108, with higher scores associated with less healthy dietary intake.
Time Frame: Baseline, 48 weeks after first group session
Population: Participants who completed the dietary risk assessment at baseline and 48 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HARMONY | Nutrition and Exercise Education Workgroup (NEEW)
Number analyzed (Participants) | 41 | 32
score on a scale | 0.45 (4.32) | 2.54 (4.31)

3. Primary Outcome: Change in Veggie Meter Score
Description: The participant's nutrition will be assessed using the veggie meter, which uses light reflectance spectroscopy to provide an estimated skin carotenoid composite score. Score ranges from 0 to 800, with higher scores associated with greater fruit and vegetable intake.
Time Frame: Baseline, 48 weeks after first group session
Population: Participants who provided Veggie meter data at at baseline and 48 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HARMONY | Nutrition and Exercise Education Workgroup (NEEW)
Number analyzed (Participants) | 47 | 39
score on a scale | 19.85 (81.85) | 9.38 (94.17)

4. Secondary Outcome: Change in BMI
Description: The participant's BMI is calculated as weight (kg) divided by the square of height (m^2).
Time Frame: Baseline, 48 weeks after first group session
Population: Participants who provided BMI data at baseline and 48 weeks.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | HARMONY | Nutrition and Exercise Education Workgroup (NEEW)
Number analyzed (Participants) | 48 | 40
kg/m^2 | -.09 (1.83) | -.56 (2.07)

5. Secondary Outcome: Change in Weight
Description: The participants weight will be measured using a digital scale.
Time Frame: Baseline, 48 weeks after first group session
Population: Participants who provided weight data at baseline and 48 weeks.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | HARMONY | Nutrition and Exercise Education Workgroup (NEEW)
Number analyzed (Participants) | 48 | 40
kg | -1 (4.54) | -2.08 (5.53)

6. Secondary Outcome: Change in Waist-to-Hip Ratio
Description: The participant's waist to hip ratio is calculated by using the mean of two waist circumference measurements divided by mean of two hip circumference measurements. Waist circumference will be measured at the midpoint between the upper iliac crest and lower costal margin in the midaxillary line. Hip circumference will be measured at the maximum width of the buttocks or gluteo-femoral fold.
Time Frame: Baseline, 48 weeks after first group session
Population: Participants who provided waist and hip measurements at baseline and 48 weeks.
Measure: Mean (Standard Deviation); unit: unitless ratio
Arm/Group | HARMONY | Nutrition and Exercise Education Workgroup (NEEW)
Number analyzed (Participants) | 48 | 38
unitless ratio | .05 (0.12) | 0 (0.09)

7. Secondary Outcome: Change in Percent Body Fat
Description: The participant's percent body fat is measured using lange skinfold calipers. The final measurement will be the mean of three measurements on the right side of the body.
Time Frame: Baseline, 48 weeks after first group session
Population: Participants who provided percent body fat data at baseline and 48 weeks.
Measure: Mean (Standard Deviation); unit: percent of total body mass
Arm/Group | HARMONY | Nutrition and Exercise Education Workgroup (NEEW)
Number analyzed (Participants) | 9 | 9
percent of total body mass | 1.23 (4.25) | -.62 (2.39)

8. Secondary Outcome: Change in Blood Pressure (Systolic)
Description: The participant's blood pressure is measured using an electronic sphygmomanometer. The final measurement will be the mean of three measurements.
Time Frame: Baseline, 48 weeks after first group session
Population: Participants who provided blood pressure data at baseline and 48 weeks.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | HARMONY | Nutrition and Exercise Education Workgroup (NEEW)
Number analyzed (Participants) | 45 | 34
mm Hg | 3.58 (15.17) | -1.44 (22.28)

9. Secondary Outcome: Change in Blood Pressure (Diastolic)
Description: as for outcome 8
Time Frame: Baseline, 48 weeks after first group session
Population: Participants who provided blood pressure at baseline and 48 weeks.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | HARMONY | Nutrition and Exercise Education Workgroup (NEEW)
Number analyzed (Participants) | 45 | 34
mm Hg | 0.29 (9.65) | -2.00 (10.37)

10. Secondary Outcome: Change in High Sensitivity C-Reactive Protein Amount
Description: The participant's high sensitivity C-reactive protein levels will be obtained via phlebotomy. C-Reactive Protein is an inflammatory biomarker, and indicative of cardiovascular risk. Data will be log-transformed, and the units will be log-(ng/mL).
Time Frame: Baseline, 48 weeks after first group session
Population: Participants who provided blood samples that were successfully assayed for CRP at baseline and 48 weeks.
Measure: Mean (Standard Deviation); unit: log(ng/mL)
Arm/Group | HARMONY | Nutrition and Exercise Education Workgroup (NEEW)
Number analyzed (Participants) | 38 | 37
log(ng/mL) | -0.784 (0.723) | -0.450 (0.860)

11. Secondary Outcome: Change in IL-6
Description: The participant's IL-6 levels will be obtained via phlebotomy. IL-6 is an inflammatory biomarker, and indicative of cardiovascular risk. Data will be log-transformed, and the units will be log-(pg/mL).
Time Frame: Baseline, 48 weeks after first group session
Population: Participants who provided blood samples that were successfully assayed for Il-6 at baseline and 48 weeks.
Measure: Mean (Standard Deviation); unit: log(pg/mL)
Arm/Group | HARMONY | Nutrition and Exercise Education Workgroup (NEEW)
Number analyzed (Participants) | 38 | 34
log(pg/mL) | 0.155 (0.670) | 0.819 (1.661)

12. Secondary Outcome: Change in Glycosylated Hemoglobin (HbA1c)
Description: Participant's glycosylated hemoglobin levels will be obtained via phlebotomy. Glycosylated hemoglobin amount is indicative of cardiovascular risk.
Time Frame: Baseline, 48 weeks after first group session
Population: Participants who provided fingerstick data at baseline and 48 weeks
Measure: Mean (Standard Deviation); unit: percent of hemoglobin
Arm/Group | HARMONY | Nutrition and Exercise Education Workgroup (NEEW)
Number analyzed (Participants) | 47 | 40
percent of hemoglobin | -.06 (0.61) | -.03 (0.44)

ADVERSE EVENTS:
Time Frame: From the time of randomization until study completion, up to 48 weeks.
Arm/Group | HARMONY | Nutrition and Exercise Education Workgroup (NEEW)
All-Cause Mortality (participants affected / at risk) | 0/87 | 0/86
Serious Adverse Events (participants affected / at risk) | 0/87 | 0/86
Other Adverse Events (participants affected / at risk) | 1/87 | 0/86
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HARMONY (N=87) | Nutrition and Exercise Education Workgroup (NEEW) (N=86)
Broken toes subsequent to prior condition (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-27): https://cdn.clinicaltrials.gov/large-docs/79/NCT04705779/Prot_SAP_001.pdf
  • Informed Consent Form (2022-05-27): https://cdn.clinicaltrials.gov/large-docs/79/NCT04705779/ICF_000.pdf